CLINICAL TRIAL: NCT05851287
Title: The Cohort Study of Eye Health of Aging People
Brief Title: The Aging Eye Cohort Study
Acronym: AECS
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, The Vice President of Zhongshan Ophthalmic Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2023KYPJ003
Record Dates: First submitted 2023-04-09; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Eye Diseases
Keywords: Elderly population; Common eye disease; Risk factor; Genetics
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — 16 mL whole blood for each subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aging is a major risk factor for many blind-causing eye diseases, e.g., glaucoma, age-related cataracts, and age-related macular degeneration. With the population aging, the impact of lifestyle changes (less time spent outdoors, increasingly sedentary lifestyles, and unhealthy eating habits) on the eye health of the elderly needs further research. This study focuses on establishing a cohort of elderly subjects with normal vision and ocular structure at baseline. The main goal is to study the risk factors for common eye diseases in Chinese elderly population while providing normal-controlled clinical and genomic data for other clinical studies on eye diseases.

ELIGIBILITY:
Inclusion criteria:

1. Be able and willing to consent to the qualification and the follow-up phases of the study;
2. Be able to undergo yearly examinations for ≥5 years;
3. Age is older than 60 years;
4. Best-corrected visual acuity of both eyes is better than 20/32;
5. Intraocular pressure (non-contact tonometer) is between 10-21 mmHg;
6. Except for mild cataracts, no other structural abnormalities of the eye are found.
7. have fundus photographs of adequate quality as assessed with a standardized protocol by the University of Wisconsin Fundus Photograph Reading Center.

Exclusion Criteria:

1. the presence of ocular disease in either eye, except for mild cataracts and ametropia;
2. previous retinal or other ocular surgical procedures (other than cataract extraction and capsulotomy);
3. a chronic requirement for any systemic or ocular medication administered for other diseases and known to be toxic to the retina or optic nerve;
4. cataract surgery within three months or capsulotomy within six weeks before the qualification visit;
5. any systemic disease with a poor 5-year survival prognosis.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The elderly population with normal visual acuity lives in Guangzhou, China.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2028-02-19 (Estimated); Study Completion 2029-02-19 (Estimated)

PRIMARY OUTCOMES:
The incidence of visual impairment at Year 1 | 1 Year
  The best corrected visual acuity is worse than 15/25.
The incidence of visual impairment at Year 2 | 2 Year
  The best corrected visual acuity is worse than 15/25.
The incidence of visual impairment at Year 3 | 3 Year
  The best corrected visual acuity is worse than 15/25.
The incidence of visual impairment at Year 4 | 4 Year
  The best corrected visual acuity is worse than 15/25.
The incidence of visual impairment at Year 5 | 5 Year
  The best corrected visual acuity is worse than 15/25.

SECONDARY OUTCOMES:
Change from Baseline Best Corrected Visual Acuity at 1 Year | 1 Year
Change from Baseline Best Corrected Visual Acuity at 2 Year | 2 Year
Change from Baseline Best Corrected Visual Acuity at 3 Year | 3 Year
Change from Baseline Best Corrected Visual Acuity at 4 Year | 4 Year
Change from Baseline Best Corrected Visual Acuity at 5 Year | 5 Year
The incidence of age-related cataract at Year 1 | 1 Year
  Presence of moderate to severe cataract in one or both eyes, graded by Lens Opacities Classification System III (LOCSIII).
The incidence of age-related cataract at Year 2 | 1 Year
  Presence of moderate to severe cataract in one or both eyes, graded by Lens Opacities Classification System III (LOCSIII).
The incidence of age-related cataract at Year 3 | 3 Year
  Presence of moderate to severe cataract in one or both eyes, graded by Lens Opacities Classification System III (LOCSIII).
The incidence of age-related cataract at Year 4 | 4 Year
  Presence of moderate to severe cataract in one or both eyes, graded by Lens Opacities Classification System III (LOCSIII).
The incidence of age-related cataract at Year 5 | 5 Year
  Presence of moderate to severe cataract in one or both eyes, graded by Lens Opacities Classification System III (LOCSIII).
The incidence of age-related macular degeneration at Year 1 | 1 Year
  The development of the neovascular form of AMD or the development of geographic atrophy that involves the center of the macula in one or both eyes.
The incidence of age-related macular degeneration at Year 2 | 2 Year
  The development of the neovascular form of AMD or the development of geographic atrophy that involves the center of the macula in one or both eyes.
The incidence of age-related macular degeneration at Year 3 | 3 Year
  The development of the neovascular form of AMD or the development of geographic atrophy that involves the center of the macula in one or both eyes.
The incidence of age-related macular degeneration at Year 4 | 4 Year
  The development of the neovascular form of AMD or the development of geographic atrophy that involves the center of the macula in one or both eyes.
The incidence of age-related macular degeneration at Year 5 | 5 Year
  The development of the neovascular form of AMD or the development of geographic atrophy that involves the center of the macula in one or both eyes.
The incidence of glaucoma at Year 1 | 1 Year
The incidence of glaucoma at Year 2 | 2 Year
The incidence of glaucoma at Year 3 | 3 Year
The incidence of glaucoma at Year 4 | 4 Year
The incidence of glaucoma at Year 5 | 5 Year
The incidence of diabetic retinopathy at Year 1 | 1 Year
The incidence of diabetic retinopathy at Year 2 | 2 Year
The incidence of diabetic retinopathy at Year 3 | 3 Year
The incidence of diabetic retinopathy at Year 4 | 4 Year
The incidence of diabetic retinopathy at Year 5 | 5 Year
The incidence of myopia-related fundus changes at Year 1 | 1 Year
The incidence of myopia-related fundus changes at Year 2 | 2 Year
The incidence of myopia-related fundus changes at Year 3 | 3 Year
The incidence of myopia-related fundus changes at Year 4 | 4 Year
The incidence of myopia-related fundus changes at Year 5 | 5 Year
Change from Baseline Self-scoring of the Visual Quality assessment scale at Year 1 | 1 Year
  Self-assessment of the visual quality will be evaluated by Visual Function index-14 (Chinese version) Questionnaire, higher scores mean a worse outcome.
Change from Baseline Self-scoring of the Visual Quality assessment scale at Year 2 | 2 Year
  Self-assessment of the visual quality will be evaluated by Visual Function index-14 (Chinese version) Questionnaire, higher scores mean a worse outcome.
Change from Baseline Self-scoring of the Visual Quality assessment scale at Year 3 | 3 Year
  Self-assessment of the visual quality will be evaluated by Visual Function index-14 (Chinese version) Questionnaire, higher scores mean a worse outcome.
Change from Baseline Self-scoring of the Visual Quality assessment scale at Year 4 | 4 Year
  Self-assessment of the visual quality will be evaluated by Visual Function index-14 (Chinese version) Questionnaire, higher scores mean a worse outcome.
Change from Baseline Self-scoring of the Visual Quality assessment scale at Year 5 | 5 Year
  Self-assessment of the visual quality will be evaluated by Visual Function index-14 (Chinese version) Questionnaire, higher scores mean a worse outcome.
Change from Baseline Self-scoring of the Quality of Life at Year 1 | 1 Year
  Self-assessment of the life quality will be evaluated by EQ-5D questionnaires, lowerer scores mean a worse outcome.
Change from Baseline Self-scoring of the Quality of Life at Year 2 | 2 Year
  Self-assessment of the life quality will be evaluated by EQ-5D questionnaires, lowerer scores mean a worse outcome.
Change from Baseline Self-scoring of the Quality of Life at Year 3 | 3 Year
  Self-assessment of the life quality will be evaluated by EQ-5D questionnaires, lowerer scores mean a worse outcome.
Change from Baseline Self-scoring of the Quality of Life at Year 4 | 4 Year
  Self-assessment of the life quality will be evaluated by EQ-5D questionnaires, lowerer scores mean a worse outcome.
Change from Baseline Self-scoring of the Quality of Life at Year 5 | 5 Year
  Self-assessment of the life quality will be evaluated by EQ-5D questionnaires, lowerer scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No